CLINICAL TRIAL: NCT05651685
Title: Assesment of TDApp2 an eHelath Tool to Make Pharmacologic and Non-pharmacologic Treatment Recommendations for Patients With ADHD
Brief Title: Treatment Recommendations for Patients With ADHD TDApp2
Status: Completed | Type: Observational
Sponsor: Universitat de Girona (Other)
Collaborators: Institut d'Assistència Sanitària (Other)
Responsible Party: Principal Investigator, Xavier Castells, Principal Investigator, Universitat de Girona
Other Study IDs: TDApp2
Record Dates: First submitted 2022-11-20; First posted 2022-12-15 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: eHealth; evidence based medicine; clinical decission support systems
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TDApp2: This cohort will use TDApp2: an eHealth tool that formulates participatory, individualized, explainatory and automated treatment recommendations for patients with Attention Deficit Hyperactivity Disorder

SUMMARY:
The purpose of this study is to compare the recommendations made by TDApp2 with those by relevant clinical practice guidelines in children/adolescents with ADHD.

DETAILED DESCRIPTION:
Clinical practice guidelines (CPG) allow optimizing medical decisions and health care based on the best evidence available. Nevertheless, CPGs have several limitations. First, many GPC are outdated shortly after their publication. Second, CPG recommendations are often not applicable to many patients treated in clinical practice. Most CPGs do not make recommendations for complex patients with comorbidities. Another limitation is that patients involvement in CPGs development is still poor. To overcome these limitations, study investigators developed TDApp, an eHealth tool to formulate decentralized, participatory, individualized and automated pharmacologic treatment recommendations for patients with Attention Deficit Hyperactivity Disorder. TDApp was initially tested in a clinical sample of ADHD patients (https://clinicaltrials.gov/ct2/show/NCT04228094), but, as it was the first human use, treatment recommendations were kept hidden to the clinicians until the last patient enrolled completed study participation. This safeguard was implemented to avoid potential misguidance. After completing this study, the investigators developed a new iteration of TDApp (TDApp2) that can also recommend non-pharmacological interventions.

In this study, the investigators aim to assess TDApp2: an eHealth tool that formulates participatory, participatory, explainatory and automated therapeutic recommendations for patients with Attention Deficit Hyperactivity Disorder. The recommendations made by TDApp2 will be compared with those made by relevant clinical practice guidelines in children/adolescents with ADHD.

A 6-week, one group, open label study will be conducted. Tirty-two children/adolescents aged < 18 yo with ADHD and their parents will use TDApp. The treatment recommendations made by the TDApp2 will be compared to those made by relevant CPG (American Academy of Pediatrics CPG, Canadian ADHD Resource Alliance (CADDRA) GPC, National Institute for Health and Care Excellence (NICE) GPC, the Australian ADHD Professionals Association guideline, and the Spanish GPC). As the study will be carried out in Catalonia (Spain), the primary comparison will be performed vs. the Spanish CPG. Also, TDApp2 recommendations will be compared with the actual treatment prescribed by the clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6-17 yo
* Meeting DSM 5 criteria for ADHD
* Requiring treatment initiation for ADHD or requiring a treatment change

Exclusion Criteria:

* Patients who are receiving treatment for ADHD and who are well controlled with it
* Patients who do not have a suitable electronic device for TDApp2

Ages: 6 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescents with ADHD requiring treatment initiation for ADHD or requiring a treatment change will be enrolled for 6 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Treatment recommended | Week 1
  Treatment recommended consists on the treatment recommended to the patient with ADHD by TDApp2 and CPG. The number and type of recommended treatments will be compared.

SECONDARY OUTCOMES:
Pharmacological distance according to the the NbN2R classification | Week 1
  The pharmacological distance corresponds to the number of pharmacological targets and modes of action that are different between two drugs according to the the NbN2R classification. E.g., the pharmacological distance between methylphenidate and atomoxetine is 16 because they are two different chemical entities and their pharmacological targets and modes of action are rather different (methylphenidates acts primarily on the dopamine (DA) neurotransmission and secondarily on the norepinephrine (NE) one, and inhibits the DA and NE transporters and releases DA and NE, while atomoxetine is a selective NE transporter inhibitor). Conversely, as methylphenidate and dexmethylphenidate act on the same pharmacological targets and have the same mode of action their pharmacological distance is 1 because they are 2 different chemical entities although closely related.
  The pharmacological distance ranges 1-26 with higher score denoting a greater pharmacological distance
ADHD symptom severity as assessed by the DSM 5 Attention-Deficit/Hyperactivity Disorder Rating Scale | Baseline and week 6
  ADHD symptom severity assessed with the DSM 5 Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS).
  The DSM 5 ADHD-RS ranges 0-54 with higher score denoting a worse outcome.
Global assessment of severity of illness as assessed by the Clinical Global Impression - Severity of Illness (CGI-S) Scale | Baseline and week 6
  The CGI-S measures symptom severity of patients with mental disorders. CGI ranges 1-7 with higher score denoting a worse outcome.
Sense of coherence as assessed by the Sense of Coherence (SOC)-13 by Antonovsky | Week 1 and week 3
  The degree to which the patient views the world and the individual environment as comprehensible, manageable, and meaningful as assessed by the Sense of Coherence (SOC)-13 by Antonovsky.
Individuals' confidence in their capacity to act in the ways necessary to reach specific goals as assessed by the Bäbler, Schwarzar, and Jerusalem self-efficacy scale | Week 1 and week 3
  The individuals' confidence in their capacity to act in the ways necessary to reach specific goals will be assessed with the Bäbler, Schwarzar, and Jerusalem self-efficacy scale.
Health literacy as assessed by the health literacy questionnaire 16-item, European Health Literacy Survey Questionnaire (HLS-EU-Q16) | Week 1 and week 3
  The degree to which individuals have the ability to find, understand, and use information and services to inform health-related decisions and actions for themselves and others. It will be assessed with the health literacy questionnaire 16-item, European Health Literacy Survey Questionnaire (HLS-EU-Q16)
Knowledge about ADHD as assessed by an ad hoc test | Week 1 and week 3
  Knowledge about ADHD will be assessed by means of an ad hoc test containing 15 statements and the patient/parent will indicate whether they are true or false. The total score ranges 0-15 with higher score denoting a better outcome.
Treatment prescribed | Week 1
  This is a qualitative outcome corresponding to the pharmacological or non-pharmacological treatment prescribed by the clinician, therfore it has no units nor range.
Patient satisfaction with the educational material as assessed by a 5-point Likert scale | Week 1
  Patients will be asked to rate their satisfaction with the educational material using a 5-point Likert scale. The total score ranges 1-5 with higher score denoting a better outcome.
Patient satisfaction with the decision-making process as assessed by a 5-point Likert scale | Week 1
  Patients will be asked to rate their satisfaction with the decision-making process using a 5-point Likert scale. The total score ranges 1-5 with higher score denoting a better outcome.
Perceived usefulness of the clinical recommendations as assessed by a 5-point Likert scale | Week 1
  Clinicians will be asked to rate the degree to which they preceive TDApp2 treatment recommendations useful using a 5-point Likert scale. The total score ranges 1-5 with higher score denoting a better outcome.
Adverse events | Weeks 3 and 6
  Adverse events occured during the study
Patient perceived satisfaction with the treatment as assessed by a 5-point Likert scale | Week 6
  Patient satisfaction with the treatment using a 5-point Likert scale. The total score ranges 1-5 with higher score denoting a better outcome.
Clinicians satisfaction with the treatment recommendations formulated by TDApp2 as assessed by a 5-point Likert scale | Week 6
  Clinician satisfaction (Clinicians fulfilment of their expectations or needs derived from the treatment recommendations formulated by TDApp2) with the treatment using a 5-point Likert scale.The total score ranges 1-5 with higher score denoting a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Castells, Principal Investigator — Universitat de Girona
Locations (1):
- Institut d'Assitència Sanitària, Salt, Catalonia, Spain